CLINICAL TRIAL: NCT06725732
Title: Assessment of Nebulized Tranexamic Acid in Functional Endoscopic Sinus Surgery Using Modena Bleeding Score. a Randomized Double Blinded Controlled Trial.
Brief Title: Assessment of Nebulized Tranexamic Acid in Functional Endoscopic Sinus Surgery Using Modena Bleeding Score
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Zanaty, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IV & Nebulized TXA in FESS
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous (Experimental)
  Interventions: Drug: Tranexamic Acid
- Nebulized (Experimental)
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — To see if nebulised TXA is better to control blood loss in functional Endoscopic sinus surgery
  Arms: Nebulized
Drug: Tranexamic Acid — To see if intravenous TXA is better to control blood loss in functional Endoscopic sinus surgery
  Arms: Intravenous

SUMMARY:
The aim of this study is to investigate the effect of preoperative administration of intravenous or nebulized tranexamic acid on surgical field, blood loss, anesthetic consumption and hemodynamics of patients undergoing FESS.

Primary outcome Modena Bleeding Score (MBS) assessing surgical field Secondary outcome

1. Patient hemodynamics.
2. Anesthetic consumption, Extra doses of fentanyl and propofol and sevoflurane>2
3. Postoperative complications: including any adverse effects to TXA e.g.nausea, vomiting, any visual disturbances, fits, and any thrombotic manifestation.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is the current standard treatment for a variety of conditions affecting the nasal cavity and the paranasal sinuses, such as chronic rhinosinusitis, benign and malignant tumors or cerebrospinal fluid leaks .Being mostly a one-handed technique, FESS does not allow simultaneous use of operative instruments and blood suction, thus endonasal bleeding control represents a challenging issue for the operating surgeon. Such narrow and highly vascularized cavities like the nasal fossae and paranasal spaces can be entirely filled with blood within few seconds, especially if the mucosa is severely inflamed as a consequence of rhinosinusitis. Bleeding is possibly the most relevant factor that could impair the quality of the surgical field during endoscopic procedures. It has been proven that uncontrolled bleeding during endoscopic sinus surgical procedures determines poor visualization of the anatomical landmarks, prolongs surgical time and carries a higher rate of complications .Several techniques to control intraoperative bleeding and improve surgical view during sinus surgery (e.g. topical vasoconstrictors, total intravenous anesthesia, controlled hypotension) have been described and analyzed to determine their efficacy .These types of studies, however, are complex and prone to bias, partially because standardized and validated methods of quantifying bleeding or grading the surgical field in endoscopic view are lacking.

Tranexamic acid functions as the competitive antagonist at the lysine site on plasminogen . During all surgical procedures, the tissue plasminogen activator is released due to tissue damage during surgery, which can convert tissue plasminogen to plasmin, promote fibrinolysis and activate the fibrinolytic system. Thus, tranexamic acid functions as an anti-fibrinolytic agent by inhibiting the tissue plasminogen activator. It can be applied topically or systemically with this mechanism in the coagulation cascade to reduce intraoperative bleeding .The results of several recent studies on endoscopic sinus surgery through topical administration of tranexamic acid are encouraging in terms of the efficacy of tranexamic acid for intraoperative bleeding and other pathological conditions .The purpose of this study is to analyze the efficacy of nebulized tranexamic acid and compare it with intravenous tranexamic acid to improve the surgeon and patient experiences of sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Either sex
2. age 18-65 years
3. ASA I-II who are listed for elective functional endoscopic sinus surgery (FESS) under general anesthesia
4. normal accepted coagulation profile and hematocrit value ≥30

Exclusion Criteria:

* • chronic renal failure

  * liver cirrhosis
  * bleeding disorders
  * current anticoagulant therapy
  * pregnancy or breastfeeding
  * impaired color vision
  * severe vascular ischemia
  * history of venous thrombosis, pulmonary embolism
  * long term treatment with acetylsalicylic acid or non-steroidal anti-inflammatory drugs not discontinued before surgery
  * hemoglobin (HB) concentration <10 mg/dl _allergy to TXA.
  * BMI > 35 kg/ m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-29 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Modena Bleeding Score- assessing surgical field | Baseline
  * No bleeding ->1.
  * Bleeding easily controlled by suctioning, washing, or packing without any significant modification or slowing of surgical procedure->2.
  * Bleeding slowing surgical procedure->3.
  * Most of the maneuvers dedicated to bleeding control ->4.
  * Bleeding that prevents every surgical procedure except those dedicated to bleeding control->5.

SECONDARY OUTCOMES:
Measuring patient's Blood Pressure-> mmhg (unit of measure) | Baseline
Measuring patient's Respiratory Rate-> breath per minute(unit of measure) | Baseline
Measuring patient's Temperature-> Celsius(unit of measure) | Baseline
Measuring patient's Pulse->Beat per minute(unit of measure) | Baseline
Measuring End-tidal Co2 by Capnogram | Baseline
  Unit of measure-> mmhg
Measuring O2 saturation by the pulse-oximeter | Baseline
Measuring amount of intraoperative bleeding through blood volume in suction jar | Baseline
Measuring the amount of intraoperative bleeding by counting gauze used in the operation. | Baseline
2. Anesthetic consumption, Extra doses of fentanyl and propofol and sevoflurane>2 | Baseline
Presence or absence of nausea as a Postoperative complication | Baseline
Presence or absence of vomiting as a Postoperative complication | Baseline
Presence or absence of any form of visual disturbance as a Postoperative complication | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Main building, Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Kang H, Hwang SH. Does topical application of tranexamic acid reduce intraoperative bleeding in sinus surgery during general anesthesia? Braz J Otorhinolaryngol. 2020 Jan-Feb;86(1):111-118. doi: 10.1016/j.bjorl.2019.08.006. Epub 2019 Oct 3. PMID 31653606
- [Background] Khosla AJ, Pernas FG, Maeso PA. Meta-analysis and literature review of techniques to achieve hemostasis in endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Jun;3(6):482-7. doi: 10.1002/alr.21126. Epub 2012 Dec 16. PMID 23255493
- [Background] Kim DH, Kim S, Kang H, Jin HJ, Hwang SH. Efficacy of tranexamic acid on operative bleeding in endoscopic sinus surgery: A meta-analysis and systematic review. Laryngoscope. 2019 Apr;129(4):800-807. doi: 10.1002/lary.27766. Epub 2018 Dec 28. PMID 30593688
- [Background] Alicandri-Ciufelli M, Pingani L, Mariano D, Anschuetz L, Molinari G, Marchioni D, Bonali M, Galeazzi GM, Presutti L. Rating surgical field quality in endoscopic ear surgery: proposal and validation of the "Modena Bleeding Score". Eur Arch Otorhinolaryngol. 2019 Feb;276(2):383-388. doi: 10.1007/s00405-018-05268-6. Epub 2019 Jan 2. PMID 30604058